CLINICAL TRIAL: NCT00127023
Title: Blinded, Randomised, Controlled Study to Evaluate the Immunogenicity and Safety of GlaxoSmithKline Biologicals' Combined Measles-mumps-rubella-varicella Candidate Vaccine Given to Healthy Children in Their Second Year of Life
Brief Title: Immunogenicity and Safety of a Combined Vaccine to Prevent Measles, Mumps, Rubella and Chickenpox Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 104389
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Mumps; Varicella; Rubella; Measles
Keywords: Prophylaxis measles, mumps, rubella and chickenpox
MeSH Terms: conditions — Mumps; Chickenpox; Rubella; Measles | interventions — Vaccines, Attenuated

INTERVENTIONS:
Biological: Measles, Mumps, Rubella and Chickenpox (live vaccine)
  Other Names: Measles; Mumps; Rubella and Chickenpox (live vaccine)

SUMMARY:
This is a study to evaluate the immunogenicity and safety of GlaxoSmithKline (GSK) Biologicals combined measles-mumps-rubella varicella candidate vaccine given to healthy children in their second year of life.

DETAILED DESCRIPTION:
Separate injections of the licensed Priorix (MMR vaccine) and Varilrix (chickenpox vaccine) serve as control.

ELIGIBILITY:
Inclusion Criteria:

* A male or female subject between 11-13 months of age (i.e. from 11 month birthday until the day before the 14 month birthday) at the time of the first vaccination.

Exclusion Criteria:

* History of previous measles, mumps, rubella and/or varicella vaccination or disease, or known exposure to any of these diseases within 30 days prior to the start of the trial
* Planned administration of a vaccine not foreseen by the study protocol from 30 days prior to each vaccination until 42-56 days after each vaccination

Ages: 11 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 944
Dates: Start 2005-05; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Antibody levels after vaccination.

SECONDARY OUTCOMES:
Safety of the study vaccines.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (69):
- Germany (69):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Bönnigheim, Baden-Wurttemberg
  - GSK Investigational Site, Bretten, Baden-Wurttemberg
  - GSK Investigational Site, Ehingen, Baden-Wurttemberg
  - GSK Investigational Site, Eppelheim, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Herbolzheim, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Kirchzarten, Baden-Wurttemberg
  - GSK Investigational Site, Ludwigsburg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Marbach, Baden-Wurttemberg
  - GSK Investigational Site, Oberkirch, Baden-Wurttemberg
  - GSK Investigational Site, Oberstenfeld, Baden-Wurttemberg
  - GSK Investigational Site, Offenburg, Baden-Wurttemberg
  - GSK Investigational Site, Pfinztal, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Tettnang, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Marktheidenfeld, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Roding, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Salzgitter, Lower Saxony
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Bützow, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Waren, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bad Oeynhausen, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Hille, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Oberhausen, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Bad Kreuznach, Rhineland-Palatinate
  - GSK Investigational Site, Bodenheim, Rhineland-Palatinate
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Gerolstein, Rhineland-Palatinate
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Bischofswerda, Saxony
  - GSK Investigational Site, Döbeln, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Stollberg, Saxony
  - GSK Investigational Site, Bredstedt, Schleswig-Holstein
  - GSK Investigational Site, Brunsbüttel, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Harrislee, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Mölln, Schleswig-Holstein
  - GSK Investigational Site, Neumünster, Schleswig-Holstein
  - GSK Investigational Site, Niebüll, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Neuhaus am Rennweg, Thuringia
  - GSK Investigational Site, Weimar, Thuringia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Schuster V, Otto W, Maurer L, Tcherepnine P, Pfletschinger U, Kindler K, Soemantri P, Walther U, Macholdt U, Douha M, Pierson P, Willems P. Immunogenicity and safety assessments after one and two doses of a refrigerator-stable tetravalent measles-mumps-rubella-varicella vaccine in healthy children during the second year of life. Pediatr Infect Dis J. 2008 Aug;27(8):724-30. doi: 10.1097/INF.0b013e318170bb22. PMID 18600190
- [Background] Schuster V et al. Immunogenicity of a Refrigerator-Stable Tetravalent MMRV Vaccine after One and Two Doses. Presented at the 24th Annual Meeting of the European Society for Paediatric Infectious Diseases (ESPID), Basel, Switzerland, 3-5 May 2006.
- [Background] Schuster V et al. Tolerability of a Refrigerator-Stable Tetravalent MMRV vaccine after One and Two Doses. Presented at the 12th International Congress on Infectious Diseases (ICID), Lisbon, Portugal, 15-18 June 2006.
- [Background] Dhillon S, Curran MP. Live attenuated measles, mumps, rubella, and varicella zoster virus vaccine (Priorix-Tetra). Paediatr Drugs. 2008;10(5):337-47. doi: 10.2165/00148581-200810050-00007. PMID 18754700
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 104389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register